CLINICAL TRIAL: NCT03935230
Title: Uncontrolled Donation After Circulatory Determination of Death (uDCDD): A Potential Solution to the Shortage of Organs in Quebec?
Brief Title: Uncontrolled Donation After Circulatory Determination of Death (uDCDD)
Acronym: uDCDD
Status: Completed | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-1416
Record Dates: First submitted 2019-04-16; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2016-06

CONDITIONS: Uncontrolled Donation After Circulatory Determination of Death
Keywords: unexpected cardiopulmonary arrest; potential organ donors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
World-wide, patients waiting for organ transplantation exceed the number of organs available. Many European countries have a uDCDD program which contribute to 10-15% of the donor pool. In Canada, this type of program does not exist. The purpose of this study is to report how many deceased person fulfill the criteria for uncontrolled DCDD in a Canadian medical center.

DETAILED DESCRIPTION:
While transplantation has become the definitive treatment for many people suffering end-stage organ failure, demand exceeds supply. For many years, donation after neurological death represented the principal source of organs for transplantation. In the last decade, prevention measures, improvements in neurocritical care, and decompressive craniectomy have led to a significant decrease in the number of non-directed donors (NDDs). In such situations, alternative sources for organ donation must be identified. Cardiac-arrest patients could provide a solution to this organ shortage. Patients who have experienced unexpected in or out of hospital cardiopulmonary arrest could become organ donors. Organ donation following uncontrolled cardiocirculatory death is currently practiced in many European countries. However, in Canada, it's not yet authorized. Yet, each deceased could save up to four lives. The purpose of this study is to determine the organ potential for a cohort of patient who had died from a cardiopulmonary arrest at the CHUS in 2015 and assess the effect of the implementation of a uDCD program on the number of additional donors.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for cardiocirculatory arrest at the CIUSSS-Estrie CHUS in 2015.

Exclusion Criteria:

* Patients with a status of no resuscitation
* Pediatric patients (<18 years old)
* Adults >65 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in one organ-donation center in Quebec that is a teaching hospital and referral center for interventional cardiology. It serves a mixed urban and rural population of 350,000.
Sampling Method: Non-Probability Sample
Enrollment: 1111 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Potential contribution of a uDCDD program on the number of additional donors. | 1 year
  Defined as (must meet all criteria):
  * Age ≤70 years old
  * Absence of obvious cause of death (rigor mortis, decapitation, overwhelming traumatic injury)
  * Absence of surgical cause of cardiac arrest
  * No sign of IV drug abuse
  * No history of malignancies

SECONDARY OUTCOMES:
Effect of the implementation of a uDCDD program on the number of additional organs suitable for transplantation. | 1 year
  Effect of the implementation of a uDCDD program on the number of additional organs suitable for transplantation.
Number of tissus donors | 1 year
  Number of tissus donors
Potential obstacles and solutions related to the implementation of a uDCDD program in Canada. | 1 year
  Potential obstacles and solutions related to the implementation of a uDCDD program in Canada.
Areas of future research. | 1 year
  Areas of future research.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérick D'Aragon, Dr/Pr, Principal Investigator — Université de Sherbrooke

IPD SHARING:
Plan to Share IPD: No